CLINICAL TRIAL: NCT01503502
Title: Phase II Study of Flumatinib Versus Imatinib in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: A Phase II Study of Flumatinib Versus Imatinib to Treat Philadelphia Chromosome Positive Chronic Myelogenous Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHGV678-201
Record Dates: First submitted 2012-01-01; First posted 2012-01-04 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Myelogenous Leukemia, Chronic
Keywords: Myelogenous Leukemia; chronce; Philadelphia Chromosome Positive; Flumatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid | interventions — flumatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- flumatinib 400mg qd (Experimental)
  Interventions: Drug: flumatinib
- flumatinib 600 mg qd (Experimental)
  Interventions: Drug: flumatinib
- imatinib (Active Comparator)
  Interventions: Drug: imatinib

INTERVENTIONS:
Drug: flumatinib — Flumatinib was supplied as 100 and 200 mg film-coated tablets for oral administration. Storage condition: 25°C, light proof, sealed.
  Other Names: HHGV678
  Arms: flumatinib 400mg qd; flumatinib 600 mg qd
Drug: imatinib — Imatinib was supplied as 100 mg film-coated tablets. Storage condition: 25°C (77°F). Protected from moisture.
  Other Names: Gleevec
  Arms: imatinib

SUMMARY:
It is an open-label, randomized, multi-center study. The efficacy and safety of two flumatinib doses, 400 mg once daily and 600 mg once daily, will be compared with imatinib 400 mg once daily in newly diagnosed (within 6 months) patients with Philadelphia chromosome-positive (Ph+) Chronic Myelogenous Leukemia in the chronic phase (CML-CP).

DETAILED DESCRIPTION:
It is an open-label, randomized, multi-center study in comparison of Gleevec and flumatinib in newly diagnosed (within 6 months) CML patients who are Philadelphia chromosome-positive. One hundred and fifty adult patients will be randomized in 1:1:1 ratio. The planned doses are as follows: 400 mg QD (50 patients) of flumatinib, 600 mg QD (50 patients) of flumatinib, and 400 mg QD (50 patients) of imatinib. Flumatinib will be dosed, based on the food effect results, in fasting condition. Imatinib will be dosed with food per the package insert. The study consists of 2 phases: 6 months of core phase and 6 months of extension phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years and ≤ 75 years of age.
2. ECOG 0, 1, or 2.
3. Diagnosis of chronic myelogenous leukemia in chronic phase with confirmation of Philadelphia chromosome.
4. Chronic myelogenous leukemia in chronic phase patients within the first 6 months of diagnosis.
5. Adequate end organ function as defined by:

   1. Total bilirubin < 1.5 x ULN,
   2. SGOT and SGPT < 2.5 x ULN,
   3. Creatinine < 1.5 x ULN,
   4. Serum amylase and lipase ≤ 1.5 x ULN,
   5. Alkaline phosphatase ≤ 2.5 x ULN unless considered tumor related.

   And patients must have the following laboratory values (≥ LLN (lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of study medication.):
   1. Potassium ≥ LLN,
   2. Magnesium ≥ LLN,
   3. Phosphorus ≥ LLN,
   4. Total calcium (corrected for serum albumin) ≥ LLN.
6. Signed informed consent.

Exclusion Criteria:

1. Previously documented T315I mutations.
2. Any medical treatment for CML prior to study entry with the exception of hydroxyurea and/or anagrelide. Treatment with tyrosine kinase inhibitor(s) prior to study entry is not allowed.
3. Treatment with other investigational agents (defined as not used in accordance with the approved indication ) within 4 weeks prior to randomization.
4. Major surgery within 4 weeks prior to randomization or who have not recovered from prior surgery.
5. Impaired cardiac function including any one of the following:

   1. History of unstable angina.
   2. History of clinically documented myocardial infarction (during the last 12 month).
   3. LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher) as determined by locally read echocardiogram.
   4. Inability to determine the QT interval on ECG.
   5. Complete left bundle branch block.
   6. Use of a ventricular-paced pacemaker.
   7. Congenital long QT syndrome or a known family history of long QT syndrome.
   8. History of or presence of clinically significant ventricular, atrial tachyarrhythmias, or QTcF > 450 msec for male or 470 msec for female.
6. Patients with active, uncontrolled psychiatric disorders including: psychosis, major depression, and bipolar disorders.
7. Severe or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection).
8. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery).
9. History of significant congenital or acquired bleeding disorder unrelated to cancer.
10. History of chronic pancreatitis or history of acute pancreatitis within 1 year of study entry.
11. Patients with another primary malignancy.
12. Acute or chronic uncontrolled liver or severe renal disease considered unrelated to disease.
13. Known to be allergic to the study drugs, including crude drug or adjuvant.
14. Patients actively receiving therapy with strong CYP3A4 inhibitors, strong CYP3A4 inducers or any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug.
15. Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test within 7 days prior to Day 1 of study and (d) female of childbearing potential unwilling to use contraceptive precautions throughout the trial (post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
To compare the rate of MMR at 6 months | 6 months
  Obtain major molecular response (MMR) rate at 6 months in newly diagnosed Ph+ CML patients through comparison of the efficacy results of flumatinib with that of imtinib.

SECONDARY OUTCOMES:
To compare the rate of MMR at 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College; Fengkui Zhang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (5):
- China (5):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Union Hospital Tongji Medical College Huazhong University of Science and technology, Wuhan, Hubei
  - The First Rffiurted Hospital of Soochow University, Suzhou, Jiangsu
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality